CLINICAL TRIAL: NCT02644772
Title: Risk Factors for Re-exacerbation After a Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Brief Title: Preventing Repeat Hospitalisations in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: INCA R-ACE
Status: Completed | Type: Observational
Sponsor: Beaumont Hospital (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor Richard W Costello, Beaumont Hospital
Other Study IDs: INCA-R-ACE
Record Dates: First submitted 2015-12-10; First posted 2016-01-01 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Acute Exacerbation of COPD; Clinical problems in COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the investigators can predict which patients are at risk of a re-exacerbation of COPD within 30 and 90 days using changes in lung capacity during the initial exacerbation.

DETAILED DESCRIPTION:
Patients admitted to hospital with an acute exacerbation of COPD will be approached to participate in the study.

The investigators will analyse changes in lung capacity (through measurement of spirometry and inspiratory capacity) and physical activity level over the first three days of admission, at discharge and at a day 30 follow-up visit. The investigators will record quality of life and symptom scores at these time points and again at a day 90 telephone visit. Data relating to the patients overall health status -disease severity, co-morbidity, cognition, psychological status, home environment and adherence to inhaled medication will be collected. The investigators will look for any relationship between these changes and a further exacerbations within 30 and 90 days.

The central hypothesis of this proposal is that the clinical course following an exacerbation of COPD may be monitored through measurement of inspiratory capacity(IC), a marker of lung hyperinflation. Resolution of an exacerbation is related to an increase in inspiratory capacity above a threshold level of improvement, after which the risk of re-exacerbation within the subsequent 30 and 90 days is low. The investigators will assess the accuracy of IC as a predictor of exacerbation and the feasibility of measuring IC during the early stages of a COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Within 72 hours of admission with an Acute Exacerbation of COPD (AE COPD) defined as "an acute change in a patient's baseline dyspnoea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in therapy" as per ATS/ERS consensus guidelines[ ] where "a change in therapy" includes the following: Prescription of antibiotics and / or systemic steroids
* Diagnosis of COPD based on GOLD criteria
* Able to give informed consent
* Willing to participate in the study

Exclusion Criteria:

* Admission reason other than AE COPD or breathlessness primarily caused by another pathology
* Already enrolled in the study
* Receiving palliative care
* Severe cognitive impairment or psychological disorder that results in inability to give informed consent or complete investigations required for the study
* Physical impairment resulting in inability to complete physiological tests

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with an acute exacerbation of COPD
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The relationship between change in inspiratory capacity(IC), from admission with an exacerbation of COPD to hospital discharge, and the risk of 30-day and 90-day re-exacerbation is reduced. | From admission to 90 days from hospitalisation with an exacerbation

SECONDARY OUTCOMES:
Relationship between changes in IC and respiratory symptoms | From admission to 30 days from hospitalisation with an exacerbation
  Medical Research Council(MRC) and Borg breathlessness scores and IC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between changes in Forced Expiratory Volume in 1 second (FEV1) and respiratory symptoms | From admission to 30 days from hospitalisation with an exacerbation
  Medical Research Council(MRC) and Borg breathlessness scores and FEV1 will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between changes in Forced Vital Capacity and respiratory symptoms | From admission to 30 days from hospitalisation with an exacerbation
  Medical Research Council(MRC) and Borg breathlessness scores and FVC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in IC and quality of life scores | From admission to 30 days from hospitalisation with an exacerbation
  COPD Assessment Test (CAT) quality of life score and IC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in FEV1 and quality of life scores | From admission to 30 days from hospitalisation with an exacerbation
  COPD Assessment Test (CAT) quality of life score and FEV1 will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in FVC and quality of life scores | From admission to 30 days from hospitalisation with an exacerbation
  COPD Assessment Test (CAT) quality of life score and FVC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in IC and gait speed | From admission to 30 days from hospitalisation with an exacerbation
  4 metre gait speed test and IC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in FEV1 and gait speed | From admission to 30 days from hospitalisation with an exacerbation
  4 metre gait speed test and FEV1 will be measured will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between change in FVC and gait speed | From admission to 30 days from hospitalisation with an exacerbation
  4 metre gait speed test and FVC will be measured at hospitalisation with an exacerbation of COPD and at 30 days post exacerbation and correlated.
Relationship between patient factors and subsequent exacerbation | 90 days from hospitalisation with an exacerbation
  The association between patient factors (to include baseline GOLD grade, Charlston co-morbidity index score, Katz index, Hospital Anxiety and Depression Scale (HADS) score, Montreal Cognitive Assessment (MOCA) score) and exacerbation in the entire cohort and in those who do and do not achieve a rise in IC compared to baseline values will be examined
Time to re-exacerbation | 90 days from hospitalisation with an exacerbation
Sensitivity of vital capacity measures taken with a bedside portable spirometer compared with those performed in the pulmonary function test laboratory | Day 3-7 of hospital admission
  Vital capacity will be measured at the bedside with a portable spirometer and using gold standard spirometry in a pulmonary function laboratory. These two measurements will then be compared and correlated.
Sensitivity of FEV1 measures taken with a bedside portable spirometer compared with those performed in the pulmonary function test laboratory | Day 3-7 of hospital admission
  FEV1 will be measured at the bedside with a portable spirometer and using gold standard spirometry in a pulmonary function laboratory. These two measurements will then be compared and correlated.
Sensitivity of inspiratory capacity (IC) measured with a bedside portable spirometer and by the gold standard body plethysmography | Day 3-7 of hospital admission
  IC will be measured at the bedside with a portable spirometer and by gold standard body plethysmography in a pulmonary function laboratory. These two measurements will then be compared and correlated.
Change in vital capacity during an exacerbation and its relationship to re-exacerbation | At days 1-3 of admission, hospital discharge and 30 days from hospitalisation with an exacerbation
Change in FEV1 during an exacerbation and its relationship to re-exacerbation | At days 1-3 of admission, hospital discharge and 30 days from hospitalisation with an exacerbation
Relationship between Exacerbation factors and re-exacerbation | 90 days from hospitalisation with an exacerbation
  The association between exacerbation severity as determined by DECAF score, need for non-invasive ventilation or critical care, length of hospital stay in the entire cohort and in those who do and do not achieve a rise in IC compared to baseline values will be examined
Relationship between Social and Environmental factors and subsequent exacerbation | 90 days from hospitalisation with an exacerbation
  The impact of patients social environment as determined by living conditions, presence of home supports, socioeconomic group in the entire cohort and in those who do and do not achieve a rise in IC compared to baseline values will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, Principal Investigator — Beaumont Hospital, Dublin, Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland